CLINICAL TRIAL: NCT01766804
Title: Effect of Bovine Colostrum on Toxicity and Inflammatory Responses During Treatment of Childhood Acute Lymphoblastic Leukaemia
Brief Title: Effect of Bovine Colostrum on Toxicity and Inflammatory Responses
Acronym: CALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steffen Husby (Other)
Collaborators: University of Southern Denmark (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Steffen Husby, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OUH-HCA-002
Record Dates: First submitted 2013-01-09; First posted 2013-01-11 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; Bovine Colostrum; Inflammation; Infection; Toxicity
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Inflammation; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization was computer based in blocks of eight to ensure an equal number of participants in each randomization group. The randomization scheme was generated by using the web site Randomization.com ⟨http://www.randomization.com⟩. The randomization center was located at the same hospital as one of the recruitment sites (OUH). The randomization list was sent directly and exclusively to the research secretariat in charge of treatment allocation. Bovine colostrum or the placebo supplement was provided in identical foil sachets differing only in randomization code. Participants, their treating physicians, and any individual involved in the coordination and implementation of the trial were masked to treatment allocation.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bovine colostrum (Experimental): A daily supplement of bovine colostrum powder.
  Interventions: Dietary Supplement: Bovine Colostrum
- Placebo (Placebo Comparator): A daily placebo supplement consisting of whole milk powder and whey protein.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Bovine Colostrum — The intervention consists of daily bovine colostrum supplementation given during the induction treatment of ALL therapy for a total of four weeks.
  Other Names: Colodan, Biodane-Pharma.
  Arms: Bovine colostrum
Dietary Supplement: placebo
  Arms: Placebo

SUMMARY:
The aim of the present study is to evaluate the ability a colostrum containing diet to limit gastrointestinal toxicity including chemotherapy induced inflammation in children treated for acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
Acute lymphoblastic leukaemia (ALL) is the most common form of childhood cancers. Cure rates are improving, but the intensity of treatment is limited by toxicity. 2-5% of patients die of treatment related complications, mostly related to therapy-induced toxicity and immune suppression. The aim of the present study is to evaluate the ability a colostrum containing diet to limit gastrointestinal toxicity including chemotherapy induced inflammation. The study is based on patients treated according to the current NOPHO protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated according to the Nordic Society of Pediatric Haematology and Oncology (NOPHO) ALL protocol

Exclusion Criteria:

* Milk Allergy
* Lactose intolerance

Ages: 1 Year to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Days with fever. Fever | Measured two times daily and on suspicion during the intervention period, up to four weeks,
  Days with temperature at or above 38.5 degrees celsius.

SECONDARY OUTCOMES:
Days in intensive care unit | During the 4 week intervention period
  Number of days treated in an intensive care unit.
Days in i.v. antibiotic treatment. | During the 4 week intervention period.
  Number of days in intravenous antibiotic treatment during the intervention period.
Duration of cytopenia (neutrocytes <1,0 and platelets <20) | During the 4 week intervention period.
Proven or suspected infections | During the 4 week intervention period
  Episodes of suspected or culture positive sepsis number of documented septic events either culture proven or those treated with a course of antibiotics.
Number of blood and platelet transfusions given during the course of treatment | During the 4 week intervention period.
  Number of blood and platelet transfusions given during the course of treatment
Clinical and paraclinical indices of gastrointestinal toxicity | At base line and weekly during the 4 week intervention period. Up to 4 weeks.
  Clinical toxicity is scored using Common Toxicity Criteria for Adverse Effects (NCI-CTCAE), WHO and oral mucositis assessment scale (OMAS) grading schemes at inclusion and weekly during the treatment period. Furthermore the patients register toxicity using the oral mucositis daily questionaire(OMDQ).
  Paraclinical indices are citruline, fecal calprotectin,
Serologic markers for systemic inflammation | Weekly and at day 3 and 24, up to 4 weeks.
  Serum will be taken weekly. Markers will include C reactive protein (CRP), procalcitonin (PCT), soluble urokinase plasminogen activator receptor (sUPAR), plasma cytokines and receptors (IL-6, IL-8, Soluble tumour necrosis factor receptors (sTNFR1), IL-1Ra).
  Cytokine production in full blood cultures will be measured at day 3 and at day 24. Initial screening for a broad spectrum of cytokines will be performed in 5-10 patients. Based on these results a final panel of analyses comprising a narrower spectrum of cytokines will be determined and used for further investigation. These will include at least TNFR1, IL-1Ra, IL-6, IL-8.

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Rathe, MD, Principal Investigator — University og Southern Denmark; Steffen Husby, MD, DMSc, Study Chair — Odense University Hospital; Klaus Müller, MD, DMSc, Study Chair — Rigshospitalet, Denmark; Peder S Wehner, MD, PhD, Study Chair — Odense University Hospital; Per T Sangild, DVSc, DMSc, Study Chair — Department of Human Nutrition, Faculty of Life Science, University of Copenhagen, Denmark
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense

REFERENCES:
- [Derived] Rathe M, De Pietri S, Wehner PS, Frandsen TL, Grell K, Schmiegelow K, Sangild PT, Husby S, Muller K. Bovine Colostrum Against Chemotherapy-Induced Gastrointestinal Toxicity in Children With Acute Lymphoblastic Leukemia: A Randomized, Double-Blind, Placebo-Controlled Trial. JPEN J Parenter Enteral Nutr. 2020 Feb;44(2):337-347. doi: 10.1002/jpen.1528. Epub 2019 Mar 12. PMID 30861163
- [Derived] Shen RL, Pontoppidan PE, Rathe M, Jiang P, Hansen CF, Buddington RK, Heegaard PM, Muller K, Sangild PT. Milk diets influence doxorubicin-induced intestinal toxicity in piglets. Am J Physiol Gastrointest Liver Physiol. 2016 Aug 1;311(2):G324-33. doi: 10.1152/ajpgi.00373.2015. Epub 2016 Jul 21. PMID 27445347